CLINICAL TRIAL: NCT02521454
Title: A Pilot Trial of Mindfulness-Based Resilience Training Among Police Officers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Responsible Party: Principal Investigator, Michael Christopher, PhD, Associate Professor, Pacific University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21AT008854-01 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Mindfulness
Keywords: policing; resilience; implicit bias; violence
MeSH Terms: conditions — Bias, Implicit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBRT (Experimental): Mindfulness-Based Resilience Training
  Interventions: Behavioral: MBRT
- WL Control (No Intervention): waitlist control group

INTERVENTIONS:
Behavioral: MBRT
  Arms: MBRT

SUMMARY:
Successful policing requires rapid and unbiased decision-making, well-developed emotion regulation skills, and psychological resilience. However, law enforcement officers (LEOs) are frequently exposed to intensive work-related stress and trauma, and consequently, are at elevated risk of adverse mental health outcomes. These mental health issues in turn are some of the primary mechanisms underlying other- and self-directed violence among LEOs. The excessive use of force by LEOs, including unjustified shootings, frequently captures national headlines and is considered by many to be one of the most serious and divisive human rights issues in the United States. Previous research suggests that LEOs can be impacted by various factors when making rapid decisions while using firearms, including a lack of careful consideration of contextual factors and unconscious racial stereotypes. This is especially true when their cognitive and emotional resources are compromised due to factors such as stress. Similarly, key precursors to suicide among LEOs include chronic stress, exposure to trauma, alcohol misuse, and depression. The substantial personal, social, and economic costs of LEO stress, including unjustified shootings and suicide, suggest a clear need for innovative and novel prevention programs to promote well-being and reduce violence. Given its demonstrated impact on many of the precursors to self- and other-directed violence among LEOs, one possible approach is an adapted Mindfulness-Based Stress-Reduction (MBSR) program, developed specifically for LEOs. Therefore, the primary objectives of this proposal are to: (1) assess the feasibility of recruitment, adherence to program intervention, and compliance with assessment instruments, and (2) determine the impact of an adapted MBSR program (Mindfulness-Based Resilience Training; MBRT) on precursors to other- and self-directed violence, and in promoting psychological resilience and emotion regulation among LEOs. There is promising preliminary evidence suggesting that mindfulness is an effective strategy for LEOs to decrease stress and its negative outcomes, enhance resilience and emotion regulation, and ultimately reduce other- and self-directed violence. The proposed project will test the impact of MBRT using a pilot feasibility randomized controlled trial (RCT). This research will generate important information on the feasibility of recruitment, adherence to program intervention, and compliance with assessment instruments, and data obtained through the proposed study will build on the investigators existing work to provide support for a larger RCT examining the efficacy of MBRT in reducing violence.

ELIGIBILITY:
Inclusion Criteria:

* full-time, active status, sworn-in law enforcement officers in the Portland Metro area

Exclusion Criteria:

* previously completed MBRT or MBSR course

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Depression Scores on the Patient Reported Outcomes Measurement Information System (PROMIS) | 6 months
Decision Making as measured by the Shooter Bias Task | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific University, Forest Grove, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We are committed to advancing knowledge in the scientific community and the role that data sharing takes in this endeavor. We commit to compliance with NIH policies regarding sharing of unique research resources and compliance with the NIH Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources (64 FR 72090, December 23, 1999). The data generated in this grant will be presented at national or international conferences and published in a timely fashion. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central.

REFERENCES:
- [Result] Christopher MS, Hunsinger M, Goerling LRJ, Bowen S, Rogers BS, Gross CR, Dapolonia E, Pruessner JC. Mindfulness-based resilience training to reduce health risk, stress reactivity, and aggression among law enforcement officers: A feasibility and preliminary efficacy trial. Psychiatry Res. 2018 Jun;264:104-115. doi: 10.1016/j.psychres.2018.03.059. Epub 2018 Mar 23. PMID 29627695
- [Derived] Christopher M, Ferry M, Simmons A, Vasquez A, Reynolds B, Grupe D. Psychometric properties of the Buss-Perry Aggression Questionnaire-short form among law enforcement officers. Aggress Behav. 2024 Mar;50(2):e22145. doi: 10.1002/ab.22145. PMID 38477412
- [Derived] Kaplan J, Bergman AL, Green K, Dapolonia E, Christopher M. Relative Impact of Mindfulness, Self-Compassion, and Psychological Flexibility on Alcohol Use and Burnout Among Law Enforcement Officers. J Altern Complement Med. 2020 Dec;26(12):1190-1194. doi: 10.1089/acm.2020.0178. Epub 2020 Oct 5. PMID 33017172